CLINICAL TRIAL: NCT04662099
Title: Safety and Efficacy of the Bispecific CAR T Therapy Targeting CS1 and BCMA in Patients With Relapsed/ Refractory Multiple Myeloma: a Single-center, Open-label, Single-arm Clinical Study
Brief Title: T Cells Expressing a Bispecific CAR Targeting CS1 and BCMA in Relapsed/Refractory Multiple Myeloma
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Collaborators: Wuhan Si'an Medical Technology Co., Ltd (Unknown)
Responsible Party: Principal Investigator, MEI HENG, Proferssor, Cheif Doctor, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CS1+BCMA bispecific CART
Record Dates: First submitted 2020-12-03; First posted 2020-12-10 (Actual); Last update posted 2023-08-16 (Actual); Status verified 2023-08

CONDITIONS: CS1+ or BCMA+ Multiple Myeloma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Conditioning chemotherapy plus CAR T cells infusion (Experimental)
  Interventions: Biological: Conditioning chemotherapy followed by CAR T cell infusion

INTERVENTIONS:
Biological: Conditioning chemotherapy followed by CAR T cell infusion — Conditioning chemotherapy: Cyclophosphamide 250 mg/m^2 and fludarabine 30 mg/m^2 IV infusion on days -5, -4, and -3 CAR T cells infusion: 0.75x10^6-3.0X10^6 CAR+ T cells per kg of recipient bodyweight. if DLTs don't occur at the dose of 3.0X10^6 CAR+ T cells per kg, the investigators will discuss whether to try higher dose.

SUMMARY:
This is a single-center, open-label, single-arm study to evaluate the safety and efficacy of the bispecific CAR T cells targeting CS1 and BCMA in patients with relapsed or refractory multiple myeloma.

DETAILED DESCRIPTION:
* Multiple myeloma(MM) is one of the most common hematological malignancies with substantial morbidity and mortality.
* In recent years, several new therapies have prolonged survival of patients with MM, but it is still an incurable malignancy of plasma cells.
* B-cell maturation antigen (BCMA) is expressed by normal and malignant plasma cells and a small subset of B cells. This specific expression pattern makes BCMA an ideal target antigen for immunotherapies in MM.
* BCMA-targeted chimeric antigen receptor (CAR) T cells have exhibited significant efficacy in MM, but relapse due to single-target escape or poor in vivo persistence has been reported.
* Dual-targets or sequential infusion have been proposed to reduce relapse and improve outcomes post BCMA-specific CAR T therapies.
* CS1 is expressed on pro-B cells and plasma cells especially malignant ones and some evidence suggests it plays a role in stromal cell interaction in the BM tumour microenvironment.
* We have constructed a bispecific CAR containing anti-CS1 single chain variable region (scFv) and an anti-BCMA scFv in 4-1BB-containing second-generation formats.
* The bispecific CAR T cells have exhibited potent cytotoxicity in various BCMA+ or/and CS1+ MM cells and can effectively eradicate MM cells in xenograft mice models.
* This study aims to evaluate prelimary safety and efficacy of the CS1&BCMA CAR T cells in patients with relapsed or refractory MM.

ELIGIBILITY:
Inclusion Criteria:

Each potential subject must meet all of the following criteria to be enrolled in the study:

1. Aged 18-78 years old, males or females.
2. Relapsed or refractory multiple myeloma according to IMWG diagnostic criteria.
3. Received at least 2 prior lines of treatment for multiple myeloma, including a proteasome inhibitor and an immunomodulatory drug.
4. Detectable MM cells in bone marrow by conventional morphologic methods or flow cytometry, and positive expression of CS1 or BCMA on MM cells as confirmed by immunohistochemistry or flow cytometry.
5. Measurable diseases at screening as defined by any of the following:

   * Serum M-protein level ≥1.0g/dL;
   * Urine M-protein level ≥200mg/24 hours;
   * Serum immunoglobulin free light chain(FLC) ≥10 mg/dL provided abnormal FLC ratio.
6. Recovery to grade 1 or baseline of toxicities due to prior treatment, excluding hematologic toxicities and toxicity of no clinical significance, like alopecia.
7. ECOG Performance Status 0 ~ 2 (ECOG status of larger than 2 points caused by MM osteolytic destruction is accepted).
8. Good organ function at screening as defined by any of the following:

   * AST and ALT ≤ 2.5×upper limit of normal (ULN);
   * Total bilirubin≤ 2.0×ULN;
   * Creatinine clearance ≥30 mL/min/1.73m2;
   * Ejection fraction of heart ≥50%, and no clinically significant abnormal ECG findings.
9. Clinical laboratory values meeting the following criteria at screening:

   * Absolute Neutrophil Count(ANC) ≥1.0×10^9/L;
   * Platelets ≥30×10^9/L;
   * Absolute Lymphocyte Count ≥1.0×10^8/L;
   * Hemoglobin(Hb) ≥6.0g/dL.
10. Women of childbearing potential must have a negative pregnancy test at screening.
11. Patients with extramedullary lesions were eligible.
12. Patients who received prior allogeneic or autologous stem cell transplantation at least three months before screening were eligible.
13. Sign the informed consent voluntarily.

Exclusion Criteria:

Any potential subject who meets any of the following criteria will be excluded from participating in the study:

1. Evidence of serious viral, bacterial, or uncontrolled systemic fungal infection.
2. Seropositive for human immunodeficiency virus (HIV) antibody.
3. Seronegative for hepatitis B antigen or a known history of hepatitis B.
4. Hepatitis C (anti-hepatitis C virus [HCV] antibody positive or HCV-RNA quantitation positive) or a known history of hepatitis C.
5. Systemic corticosteroid therapy of greater than 5 mg/day of prednisone or equivalent dose within 2 weeks prior to apheresis.
6. Active autoimmune disease or a history of autoimmune disease within 3 years.
7. The following cardiac conditions: Myocardial infarction or coronary artery bypass graft ≤6 months prior to enrollment; History of clinically significant ventricular arrhythmia or unexplained; New York Heart Association stage III or IV congestive heart failure.
8. A history of epilepsy or other central nervous system diseases or altered mental status.
9. Known life-threatening allergies, hypersensitivity, or intolerance to CAR-T cells or relevant lymphodepleting regimens (cyclophosphamide and fludarabine).
10. Pregnant or breast-feeding, or planning to become pregnant while enrolled in this study or within one year after receiving study treatment.
11. Any uncontrolled diseases, other than multiple myeloma, that may lead to abnormal death.
12. Being participating in other intervention studies.
13. Other cases excluded by the Investigators.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2020-03-25 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-related Adverse Events | within 2 years after infusion
  Therapy-related adverse events will be recorded and assessed according to the National Cancer Institute's Common Terminology Criteria for Adverse Events (CTCAE, Version 5.0).

SECONDARY OUTCOMES:
Overall response rate(ORR) and complete response rate(CRR) of administering T cells Expressing a bispecific CAR Targeting CS1 and BCMA in Relapsed/Refractory Multiple Myeloma | 2 years after infusion
  OR and CRR will be assessed from CAR T cell infusion to death or last follow-up (censored).
Overall survival(OS), duration of Response(DOR), progress-free survival(PFS) of administering T cells Expressing a bispecific CAR Targeting CS1 and BCMA in Relapsed/Refractory Multiple Myeloma | 2 years after infusion
  OS, PFS and DOR will be assessed from CAR T cell infusion to death or last follow-up (censored).

OTHER OUTCOMES:
In vivo expansion and survival of CS1&BCMA bispecific CAR T cells | 2 years after infusion
  In vivo (bone marrow and peripheral blood) rate and quantity will be determined by using flow cytometry and qPCR.

CONTACTS AND LOCATIONS:
Overall Officials: Heng Mei, M.D., Ph.D, Principal Investigator — Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Locations (1):
- Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zah E, Nam E, Bhuvan V, Tran U, Ji BY, Gosliner SB, Wang X, Brown CE, Chen YY. Systematically optimized BCMA/CS1 bispecific CAR-T cells robustly control heterogeneous multiple myeloma. Nat Commun. 2020 May 8;11(1):2283. doi: 10.1038/s41467-020-16160-5. PMID 32385241
- [Background] Mikkilineni L, Kochenderfer JN. CAR T cell therapies for patients with multiple myeloma. Nat Rev Clin Oncol. 2021 Feb;18(2):71-84. doi: 10.1038/s41571-020-0427-6. Epub 2020 Sep 25. PMID 32978608
- [Derived] Li C, Xu J, Luo W, Liao D, Xie W, Wei Q, Zhang Y, Wang X, Wu Z, Kang Y, Zheng J, Xiong W, Deng J, Hu Y, Mei H. Bispecific CS1-BCMA CAR-T cells are clinically active in relapsed or refractory multiple myeloma. Leukemia. 2024 Jan;38(1):149-159. doi: 10.1038/s41375-023-02065-x. Epub 2023 Oct 17. PMID 37848634